CLINICAL TRIAL: NCT05720377
Title: Evaluation of Exercise Application Technology and Continuous Glucose Monitoring to Improve Weight Loss and Metabolic Markers in Adolescents
Brief Title: Evaluation of Exercise Application Technology in Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Christy Foster, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007608
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; PreDiabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Obesity

STUDY DESIGN:
Intervention Model Description: longitudinal
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Obese, receives access to exercise phone application (Experimental): obese, receives access to exercise phone application and interval contact by health provider in between clinic visits , receives continuous glucose monitor
  Interventions: Device: continuous glucose monitor (Freestyle Libre
- Obese, no intervention (No Intervention): obese, receives continuous glucose monitor
- Prediabetes, receives access to exercise phone application (Experimental): prediabetes receives access to exercise phone application and interval contact by health provider in between clinic visit, receives continuous glucose monitor
  Interventions: Device: continuous glucose monitor (Freestyle Libre
- Prediabetes, no intervention (No Intervention): prediabetes, receives continuous glucose monitor
- Type 2 diabetes, receives access to exercise phone application (Experimental): prediabetes receives access to exercise phone application and interval contact by health provider in between clinic visit, receives continuous glucose monitor
  Interventions: Device: continuous glucose monitor (Freestyle Libre
- Type 2 diabetes, no intervention (No Intervention): Type 2 diabetes, receives continuous glucose monitor

INTERVENTIONS:
Device: continuous glucose monitor (Freestyle Libre — 15 minute phone interview by health care provider to assess health goals set at clinic visits.
  Other Names: Contact by health care provider
  Arms: Obese, receives access to exercise phone application; Prediabetes, receives access to exercise phone application; Type 2 diabetes, receives access to exercise phone application

SUMMARY:
The purpose of the study is to evaluate the use of an exercise phone application and a continuous glucose monitor and their impact on metabolic disease in adolescents with obesity, prediabetes and Type 2 diabetes. Participants will be asked to wear a continuous glucose monitor (Freestyle Libre) and if they are in the intervention group also participate in using an exercise phone application as well as have scheduled interval contact with a health professional in between scheduled clinic visits to assess how they are reaching their goals.

DETAILED DESCRIPTION:
Patients will be recruited directly from the Childrens of Alabama pediatric endocrine clinic. Thirty patients who have obesity, prediabetes or Type 2 diabetes will be enrolled. During the enrollment phase, flyers will be posted in clinic and emails will be distributed to potential participants. Our study team will approach interested participants during their routine clinic visit. Consent will be obtained by study team during their endocrine clinic visit. Review of their medical records will be done and age, gender and race will be extracted from the medical record. A baseline visit with vital signs, blood work, a physical exam and nutritional counseling will be completed. Once enrolled, the patients will then be randomized.Within this pilot trial, we will randomize 15 adolescents/teenagers who either have obesity, prediabetes or Type 2 diabetes, to access to an exercise regimen and 15 adolescents to control intervention using a permuted block randomization scheme. The randomization scheme will contain 6 blocks of size 5 allowing for 30 randomized in the group with obesity, prediabetes and Type 2 diabetes.

Those who are in the intervention group will then be given access to frequent telephone counseling to follow-up their nutrition and exercise goals, access to exercise application and accelerometer as described below. Follow-up will then be completed at 3 and 6 months with a physical exam, vital signs, blood draw.

Intervention Group

Access provided to exercise application Provided with Fitbit to wear and measure activity Weekly check-in with provider to determine how exercise goals have been that week. If unable to reach, we will text securely a clinic check-in and provide a healthy tip of the week.

Meeting with nutrition at Baseline visit

Continuous glucose monitor provided (plan to wear for 14 days during each month)

Non-Intervention Group

Meeting with nutrition at Baseline visit

Continuous glucose monitor provided (plan to wear for 14 days at baseline visit, 3 month visit and 6 month visit)

ELIGIBILITY:
Inclusion Criteria for Type 2 diabetes arm

* BMI > 95th percentile
* A1c> 6.5%
* Age 14-17 (2 years post-menarchal)

Inclusion for Prediabetes Arm

* Age 14-17 (2 years post-menarchal)
* A1c 5.7-6.4%

Inclusion for Obesity Arm

* Age 14-17 (2 years post-menarchal)
* A1c 5.7-6.4%

Exclusion Criteria for all arms

* BMI <95th percentile
* Specific obesity syndrome
* Inability to participate in exercise workouts

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
skin fold thickness | baseline
  reliable estimate of subcutaneous fat at various sites of the body
skin fold measurement | 3 month
  reliable estimate of subcutaneous fat at various sites of the body
skin fold measurement | 6 month
  reliable estimate of subcutaneous fat at various sites of the body
Body mass index | baseline
  measure of body fat based on height and weight
Body mass index | 3 month
  measure of body fat based on height and weight
Body Mass Index | 6 month
  measure of body fat based on height and weight

SECONDARY OUTCOMES:
TNF-alpha | baseline
  inflammatory marker in the blood
TNF-alpha | 3 months
  inflammatory marker in the blood
TNF-alpha | 6 months
  inflammatory marker in the blood
IL-6 | Baseline
  inflammatory marker in the blood
IL-6 | 3 months
  inflammatory marker in the blood
IL-6 | 6 months
  inflammatory marker in the blood

IPD SHARING:
Plan to Share IPD: Yes